CLINICAL TRIAL: NCT07143812
Title: Clinical Research of Suicide Gene Expressing Allogenic Bone Marrow Derived Mesenchymal Stem Cells(MSC11FCD) in Patients With Newly Diagnosed Glioblastoma
Brief Title: A Study to Evaluate the Safety of a Stem Cell-Based Gene and Cell Therapy in Patients With Newly Diagnosed Glioblastoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CHA University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC11FCD
Record Dates: First submitted 2025-08-04; First posted 2025-08-27 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma (GBM); Newly Diagnosed Glioblastoma Multiforme
Keywords: Glioblastoma; mesenchymal stem cell; gene therapy; suicide gene
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The investigational drug into the Intratumoral administration (Other): The investigational drug in the amount of 1x10^7, 3x10^7cells per dose into the tumor or the tumor removal site using a syringe during surgery
  Interventions: Drug: MSC11FCD

INTERVENTIONS:
Drug: MSC11FCD — Administration period: Single dose Route of administration: Intratumoral administration Dose: 1x10^7, 3x10^7cells/dose Summary: Administer the investigational drug in the amount of 1x10^7, 3x10^7cells per dose into the tumor or the tumor removal site using a syringe during surgery.

SUMMARY:
This is a phase I clinical trial evaluating the safety, tolerability, and maximum tolerated dose of MSC11FCD, an investigational allogeneic bone marrow-derived mesenchymal stem cell therapy expressing a suicide gene, in patients with newly diagnosed glioblastoma. The investigational product is administered intratumorally following surgical resection. This study aims to explore whether MSC11FCD can provide a targeted, localized treatment option during the postsurgical period, potentially addressing residual tumor cells and reducing early recurrence.

DETAILED DESCRIPTION:
Glioblastoma is a highly aggressive and rapidly progressing malignant brain tumor classified as a grade IV glioma. Despite the current standard of care, including surgical resection, radiation therapy, chemotherapy, and tumor treating fields, prognosis remains poor due to high recurrence rates, tumor heterogeneity, treatment resistance, and limited drug penetration across the blood-brain barrier. Moreover, glioblastoma often exhibits rapid tumor regrowth during the postsurgical recovery period when few therapeutic options are available.

This study investigates MSC11FCD, an investigational allogeneic bone marrow-derived mesenchymal stem cell product genetically modified to express a suicide gene. The product is administered intratumorally in newly diagnosed glioblastoma patients following surgical resection. The primary objective of the study is to evaluate the safety, tolerability, and maximum tolerated dose of MSC11FCD. Secondary objectives include the assessment of preliminary efficacy signals. The study aims to explore the potential of this novel therapeutic approach to selectively target residual tumor cells and potentially delay or prevent early recurrence, thereby contributing to improved patient outcomes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 to 70
* Patients diagnosed with newly diagnosed glioblastoma based on medical imaging after receiving standard therapy for glioblastoma
* Patients whose expected survival period is at least 3 months
* Patients who have not received any other types of immunotherapy
* Patients who have been given a sufficient explanation of the purpose and details of the clinical trial and the characteristics of the investigational drug from an investigator and who signed the consent form or had a legal guardian or representative sign the consent form prior to the beginning of this clinical trial

Exclusion Criteria:

* Patients with recurrent glioblastoma. Known Dihydropyrimidine Dehydrogenase (DPD) deficiency Contraindications to contrast-enhanced MRI (e.g., patients with pacemakers or other reasons preventing MRI scans according to the study schedule)
* Patients who received Gliadel wafer implantation during surgery
* Patients with severe dysfunction of major organs (liver, kidney, bone marrow, lung, heart) as determined by the investigator
* Patients with concurrent malignancies other than glioblastoma or a history of malignancy within the past 5 years
* Patients with uncontrolled hypotension or hypertension
* Patients with serious infections as determined by the investigator, including sepsis, hepatitis A, B, or C
* Patients with a Karnofsky Performance Scale (KPS) score < 50
* Patients with autoimmune diseases involving the central nervous system (e.g., multiple sclerosis, myasthenia gravis, acute disseminated encephalomyelitis)
* Patients with a history of allergy to flucytosine (5-FC), its excipients, or 5-fluorouracil (5-FU)
* Pregnant or breastfeeding women, patients planning to become pregnant during the study period, or those unwilling to use appropriate contraception
* Participation in another clinical trial within 30 days prior to enrollment
* Any condition that, in the opinion of the investigator, would make the patient unsuitable for study participation

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number Of Adverse Events related to the treatment | Up to 12 months after treatment administration (Day 0)
  Evaluate the number of adverse event related to the treatment according to CTCAE V4.0 during the trial (including clinically significant changes in physical examination, radiographic images, safety lab tests, vital signs)

CONTACTS AND LOCATIONS:
Overall Officials: Jaejoon Lim, PhD, Principal Investigator — CHA University
Locations (1):
- Bundang CHA Medical Center, Seongnam, Kyunggido, South Korea

IPD SHARING:
Plan to Share IPD: No